CLINICAL TRIAL: NCT06953557
Title: Evaluation of the Salivary-free Amino Acids Levels With Caries Activity
Brief Title: Evaluation of the Salivary-free Amino Acids Levels (Glycine , Proline , Lysine , and Alanine ) With Caries Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Abeer Ibrahim Mohammed, Princible investigator, Al-Mustansiriyah University
Other Study IDs: Mustansiriyah
Record Dates: First submitted 2025-04-15; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries
Keywords: Salivary -free amino acid measurment
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: To compare the effect of salivary glycine , proline , lysine and alanine concentration between participants with high caries activity and participants with negative caries activity — The investigators will measure Salivary-free amino acids by using reverse phase high performance liquid chromatography

SUMMARY:
This study will be aimed to investigated the correlation between levels of salivary amino acids (glycine , proline , lysine , alanine ) in the saliva of healthy children with and without active carious lesions and to estimate the predictive capacity of caries susceptibility

DETAILED DESCRIPTION:
80 healthy children (8-10 years old) will be recruited from primary schools of Baghdad city/ Iraq, will be classified according to their level of caries activity (high caries activity, n = 40; negative caries activity, n = 40). Total stimulated and unstimulated saliva will be collected to estimate the caries activity by using the Snyder test, and Amino acid analysis of the saliva will be performed by reversed phase - high performance liquid chromatography (RP-HPLC), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Children aged (8,9,10) years with different caries
* Absence of signs of gingivitis or periodontal disease.

Exclusion Criteria:

* Children out the range of age
* Children with any systemic discases.
* Children with appliances in the mouth.
* Children with appliances in the mouth.
* Children with antibiotic treatment or any other drug over the last two weeks. B

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in both genders in 8-10 years old
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Salivary-free amino acid analysis | Baseline :unstimulated saliva collection for salivary glycine , proline , lysine and alanine measurement
  Unstimulated saliva collection for salivary free amino acids analysis

IPD SHARING:
Plan to Share IPD: No